CLINICAL TRIAL: NCT02295111
Title: The BMEA Study: The Impact of Meridian Balanced Method (BM) Electro-acupuncture (EA) Treatment on Women With Chronic Pelvic Pain (CPP): A Three-arm Randomized Controlled Pilot Study.
Brief Title: Electro-acupuncture (EA) and Chronic Pelvic Pain (CPP)
Acronym: BMEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/SS/1022
Record Dates: First submitted 2014-09-23; First posted 2014-11-20 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Pain
Keywords: electro-acupuncture; chronic pelvic pain; patient practitioner interactions; TCM health consultation; meridian balanced method acupuncture
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- EA treatment and TCM health consult (Active Comparator): Participants randomized to the EA treatment will receive 2 EA +TCM health consult once a week x 4 weeks (8 total)
  Interventions: Device: EA treatment
- TCM health consult (Experimental): Participants randomized to TCM health consult will receive 2 TCM health consult once a week x 4 weeks ( 8 total)
  Interventions: Behavioral: TCM health consult
- Usual care (Active Comparator): Participants randomized to usual care will continue with their usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: EA treatment — Electro acupuncture and traditional Chinese Medicine Health consult
  Arms: EA treatment and TCM health consult
Behavioral: TCM health consult — Traditional Chinese Medicine Health Consult without needling
  Arms: TCM health consult
Other: Usual Care — Standard NHS care
  Arms: Usual care

SUMMARY:
Chronic pelvic pain (CPP) is a debilitating condition that affects over 1 million women in the United Kingdom. The annual healthcare costs are estimated at over £150 million. Proven interventions which include the use of analgesics or hormonal treatments are unsatisfactory in many cases.

The investigators believe that the meridian balance method (BM) electro-acupuncture (EA) treatment (which includes a Traditional Chinese Medicine Health Consultation [TCM HC]) may be helpful in the management of CPP. Studies on the mechanisms of EA have demonstrated an analgesic effect. A recent individual patient data meta-analysis on the use of acupuncture for four chronic pain conditions found a small statistically significant effect size when compared to sham acupuncture. The effect size was larger and statistically significant when compared to usual care controls. This meta-analysis, and other large studies, suggests that, in addition to this analgesic effect, the interaction between the patient and the healthcare provider also plays a role in its effect on painful symptoms.

Our hypothesis is that the meridian BMEA treatment alleviates pain, and improves physical and emotional functioning, in women with CPP.

The investigators plan to undertake a single centre pilot study to assess the feasibility of performing a future three-armed randomised controlled, parallel group design trial to determine the efficacy of the meridian balance method electro-acupuncture (BMEA) treatment in the management of women with CPP.

The primary objective is to determine whether it is possible to achieve acceptable recruitment and retention rates within defined inclusion/exclusion criteria.

The secondary objectives are to determine the effectiveness and acceptability to patients of the proposed methods of recruitment, randomisation, interventions and assessment tools.

The investigators aim to recruit 30 women with CPP in NHS Lothian over a 12-month period and randomise them to BMEA treatment, TCM HC or standard care (SC). Response to the intervention will be monitored by validated pain, physical and emotional functioning questionnaires at weeks 0 (baseline), 4 (end of study) 8 and 12. Focus group discussion to gain feedback on study experience will be conducted at the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pelvic pain longer than 6 months duration
* Average numerical pain score of at least 4 out of 10 in the previous week
* Able and willing to comply with intervention
* Women aged 18 and above

Exclusion Criteria:

* Pregnancy
* Malignancy
* Severe bleeding disorders (e.g. Type 2, 3 Von Willebrand disease)
* Severe needle phobia
* Taking anti-coagulants
* A history of seizure
* A pace-maker in situ
* Moderate to severe psychiatric illness (currently under the care of a psychiatrist)
* Had received electro-acupuncture and meridian balanced method within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine whether it is possible to achieve acceptable recruitment and retention rates within defined inclusion/exclusion criteria. | At the end of study: 12 months from start of study
  We aim to recruit 30 women with CPP in NHS Lothian over a 12-month period and randomise them to BMEA treatment, TCM HC or standard care (SC). Response to the intervention will be monitored by validated pain, physical and emotional functioning questionnaires at weeks 0 (baseline), 4 (end of study) 8 and 12. Focus group discussion to gain feedback on study experience will be conducted at the completion of the study.

SECONDARY OUTCOMES:
The secondary objectives are to determine the effectiveness and acceptability to patients of the proposed methods of recruitment, randomisation, interventions and assessment tools. | 12 months from date of recruitment
  We aim to recruit 30 women with CPP in NHS Lothian over a 12-month period and randomise them to BMEA treatment, TCM HC or standard care (SC). Response to the intervention will be monitored by validated pain, physical and emotional functioning questionnaires at weeks 0 (baseline), 4 (end of study) 8 and 12. Focus group discussion to gain feedback on study experience will be conducted at the completion of the study.
VAS Scale | At 0, 4, 8, 12 weeks
  Questionnaire
Brief Pain Inventory | At 0, 4, 8, 12 weeks
  Questionnaire
Hospital Anxiety and Depression Scale | at 0, 4, 8, 12 weeks
  Questionnaire
SF 12 | at 0, 4, 8, 12 weeks
  Questionnaire
Work Productivity & Activity Impairment Questionnaire | at 0, 4, 8, 12 weeks
  Questionnaire
Sexual Activity Questionnaire | at 0, 4, 8, 12 weeks
  Questionnaire
Pain Catastrophising Questionnaire | at 0, 4, 8, 12 weeks
  Questionnaire
Focus Group Discussions | At the end of study
  Qualitative Method

CONTACTS AND LOCATIONS:
Overall Officials: Marie Fallon, MD PhD, Principal Investigator — University of University
Locations (1):
- Ooi Thye Chong, Edinburgh, City of Edinburgh, United Kingdom

REFERENCES:
- [Derived] Chong OT, Critchley HO, Horne AW, Elton R, Haraldsdottir E, Fallon M. The BMEA study: the impact of meridian balanced method electroacupuncture on women with chronic pelvic pain-a three-arm randomised controlled pilot study using a mixed-methods approach. BMJ Open. 2015 Nov 17;5(11):e008621. doi: 10.1136/bmjopen-2015-008621. PMID 26576808